CLINICAL TRIAL: NCT01941966
Title: A Phase II Study of Substitution of 5-FU (Fluorouracil) by Capecitabine in Scheme of Chemo-radiotherapy in Patients With Squamous Cell Carcinoma of the Anal Canal.
Brief Title: A Study of Substitution of 5-FU (Fluorouracil) by Capecitabine in Scheme of Chemo-radiotherapy in Patients With Squamous Cell Carcinoma of the Anal Canal.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP 84/2010
Record Dates: First submitted 2013-09-05; First posted 2013-09-13 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Anal Canal Cancer.
Keywords: Anal canal cancer;capecitabine; mitomycin; radiotherapy.
MeSH Terms: conditions — Anal Canal Carcinoma | interventions — Capecitabine; Mitomycins; Radiotherapy

ARMS (1):
- Chemo-radiotherapy (Experimental): Capecitabine, PO, 825mg/m2 Mitomycin C, IV, 15 mg/m2 Radiotherapy - 50,4 - 54 Gy
  Interventions: Drug: Capecitabine; Drug: Mitomycins; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Capecitabine — Capecitabine, PO, 825mg/m2, on days: 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15, 16, 17, 18, 19, 22, 23, 24, 25, 26, 29, 30, 31, 32, 33, 36, 37, 38, 39 and 40 of radiotherapy period.
Drug: Mitomycins — 15 mg/m2, IV, bolus, single dose on day 1 of radiotherapy
Radiation: Radiotherapy — Dose: 50,4-54 Gy 28 to 30 fractions during 5 to 6 weeks

SUMMARY:
The squamous cell carcinoma (SCC) of the anal canal is an uncommon neoplasia which corresponds to 1-5% of intestinal tumors. However the risk of SCC of the anal canal has been growing recently. The standard treatment of anal cancer stage II-III is multimodal and consists of combined chemotherapy (infusional 5-fluorouracil and mitomycin) and radiotherapy. This scheme currently used was proposed in 1974, and since then no other effective treatment has been developed.

The purpose of this study is to determine the efficacy and toxicity of the combination of capecitabine and mitomycin with radiotherapy in patients with carcinoma of the anal canal. For this will be selected 51 patients to be treated with chemo-radiotherapy.

The primary endpoint will be local control rate after 6 months of the end of radiotherapy and chemotherapy, defined by the rate of radiological and clinical neoplasia.

ELIGIBILITY:
Inclusion Criteria:

* Invasive anal canal SCC histologically confirmed, T2-4 N0 M0, T (anyone) N1-3 M0 - according to TNM staging system.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2.
* Adequate medullar function, defined as: Absolute neutrophil count ≥ 1,5×109/L; platelets ≥100×109/L; hemoglobin ≥10g/dl.
* Serum AST (aspartato aminotransferase) and ALT (alanine aminotransferase) < 3 × ULN (upper limit of normal).
* Serum Creatinine ≤ 1,5 ULN and clearance of creatinine estimated (Cockcroft- Gault) ≥ 50 ml/min.
* Signed written informed consent.

Exclusion Criteria:

* Major surgical procedure within 4 weeks of the beginning of the treatment.
* History of severe systemic or psychiatric disease.
* Previous treatment for anal canal carcinoma or other cancer.
* For female patients, current pregnancy and/or lactation
* Unstable angina or acute myocardial infarction within 6 months.
* Concomitant use of oral anticoagulants
* HIV positive with result of CD4 ≤ 200.
* Previously pelvic radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be local control rate after 6 months of the end of radiotherapy and chemotherapy, defined by the rate of radiological and clinical neoplasia. | 6 months of the end of radiotherapy and chemotherapy.

SECONDARY OUTCOMES:
Treatment Toxicity | Weekly during the treatment and ultil 28 days after the last dose of capecitabine or ultil the resolution of all adverse events.
  Adverse events grade 3 and 4 according to CTCAE 3.0 (Common Toxicity Criteria for Adverse Effects).
Complete Response | 4 weeks after the end of the treatment
  Complete response rate 4 weeks after completion of chemotherapy and radiation therapy.
Overall survival | Every 3 months during the first year after the end of the treatment, then every 6 months in the second and third year, and after the fourth year the visit will be annual.
Progression-free survival | A chest x-ray and computerized tomography of abdomen and pelviswill be performed after 6 weeks of the end of treatment and 6 months after.
Colostomy rate | Within 1 year after the end of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo MG Hoff, PHD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- ICESP, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Related Info — http://www.icesp.org.br